CLINICAL TRIAL: NCT03292783
Title: An Open-label, Dose-escalation and Expansion Phase 1/2a Clinical Trial to Assess the Tolerability, Safety, Pharmacokinetics, Pharmacodynamics and the Anti-tumor Efficacy of NOV1501 (ABL001) in Patients With Advanced Solid Tumors
Brief Title: This is a Study to Evaluate the Safety and Tolerability of the Study Drug ABL001, and to Determine the Maximum Tolerated Dose and/or Recommended Phase 2 Study Dose of ABL001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ABL Bio, Inc. (Industry)
Collaborators: National OncoVenture (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NOV150101-101
Record Dates: First submitted 2017-09-21; First posted 2017-09-26 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Advanced Solid Tumors
Keywords: VEGF; DLL4; Solid Tumors; bispecific antibody; anti-angiogenic
MeSH Terms: interventions — asciminib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NOV150101 (ABL001) (Experimental)
  Interventions: Drug: NOV1501 (ABL001)

INTERVENTIONS:
Drug: NOV1501 (ABL001) — VEGF/DLL4 targeting bispecific antibody

SUMMARY:
The purpose of this open-label, dose escalation-dose expansion, Phase 1 clinical trial is to evaluate the safety, pharmacokinetics and anti-tumor activity and determine the maximum tolerated dose (MTD) and recommended phase II dose (RP2D) of NOV1501 (ABL001).

DETAILED DESCRIPTION:
This is an open-label, Phase 1 dose escalation and expansion study of NOV1501 (ABL001) to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics and the anti-tumor efficacy of ABL001 in patients with advanced solid tumors after failure of standard of care.

Patients will be enrolled in two stages: a dose-escalation stage and an expansion phase. DLTs will be assessed as the primary endpoint in this trial.

ELIGIBILITY:
Inclusion Criteria:

* ≥19 year old patients with histologically or cytologically confirmed metastatic or unresectable advanced solid tumors
* Lesions measured by tumor markers or by CT/MRI must be evaluable based on response evaluation criteria in solid tumors (RECIST) version 1.1.
* Life expectancy ≥12 weeks
* ECOG performance status ≤2
* Women of childbearing potential must have a negative pregnancy test outcome
* Patients must provide written informed consent to voluntary participation in this study.

Exclusion Criteria:

* History of hypersensitivity reactions to any of the components of the investigational product or other drugs of the same class
* Less than 4 weeks have elapsed since a major surgery and 2 weeks have elapsed since a minor surgery
* New York Heart Association (NYHA) class ≥II congestive heart failure (CHF)
* Persistent, clinically significant NCI-CTCAE v4.03 Grade ≥2 toxicities from the previous anticancer therapy
* Severe infections or severe traumatic systemic disorders
* Symptomatic or uncontrolled central nervous system (CNS) metastasis
* Pregnant or lactating women or patients planning to become pregnant during the study
* Participation in another clinical trial within 30 days prior to screening
* Administration of antiplatelets or anticoagulants within 2 weeks prior to screening
* Requiring continuous treatment with systemic NSAIDs or systemic corticosteroids
* HIV or other severe diseases that warrant the exclusion from this study
* Peritoneal and/or pleural fluid drainage within 28 days prior to screening
* History of hemoptysis within 28 days prior to screening
* Serious, untreated scar, active ulcer, or untreated fracture

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2021-03-02 (Actual); Study Completion 2021-03-02 (Actual)

PRIMARY OUTCOMES:
Number and percentage of subjects with adverse events (AEs), serious adverse events (SAEs), and dose-limiting toxicities (DLTs) | From time of 1st administration of ABL001 until day 21.
  The maximum tolerated dose/maximum administered dose will be determined by the number of participant experiencing DLTs. The safety profile will be assessed through number of participants experiencing AEs, SAEs, abnormal laboratory parameters, vital signs and electrocardiogram (ECG) results.

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam-si
  - Samsung Medical Center, Seoul

REFERENCES:
- [Derived] Yeom DH, Lee YS, Ryu I, Lee S, Sung B, Lee HB, Kim D, Ahn JH, Ha E, Choi YS, Lee SH, You WK. ABL001, a Bispecific Antibody Targeting VEGF and DLL4, with Chemotherapy, Synergistically Inhibits Tumor Progression in Xenograft Models. Int J Mol Sci. 2020 Dec 29;22(1):241. doi: 10.3390/ijms22010241. PMID 33383646